CLINICAL TRIAL: NCT02524392
Title: Effect Evaluation of Independent Medical Evaluation (IME) After Six Months Sick Leave: A Randomized Controlled Trial of Independent Medical Evaluation (IME) Versus Treatment as Usual in Norway
Brief Title: Effect Evaluation of Independent Medical Evaluation (IME) in Norway
Acronym: NIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: Norwegian Labour and Welfare Administration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UniResearch
Record Dates: First submitted 2015-06-23; First posted 2015-08-14 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: All International Classification of Primary Care 2 Diagnoses
Keywords: independent medical evaluation; sick leave; sickness absence; physician primary care; general practitioner; family physician
MeSH Terms: interventions — Independent Medical Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Independent medical evaluation (Experimental): Independent medical evaluation (IME) of another doctor than the treating general practitioner.
  Interventions: Other: Independent medical evaluation
- Treatment as usual (No Intervention): Treatment as usual by the treating general practitioner. There will be one randomized control group in one county. Sick-listed in other counties serve as an extra control group.

INTERVENTIONS:
Other: Independent medical evaluation — The independent medical evaluation (IME) will be performed by specialists in general medicine, temporarily hired by the county welfare service. The independent medical evaluation (IME) procedure is developed by the Research Unit for General Practice at Uni Research Health in Norway.
  Arms: Independent medical evaluation

SUMMARY:
A randomized controlled trial comparing independent medical evaluation (IME) to treatment as usual (TAU). Participants will be individuals reaching six months uninterrupted sickness absence. Treatment as usual (TAU) is normal follow-up by a general practitioner (GP).

DETAILED DESCRIPTION:
A randomized controlled trial in a Norwegian context, involving an effect evaluation, a cost-benefit evaluation and a qualitative evaluation. Independent medical evaluation (IME) will be compared to treatment as usual (TAU). Independent medical evaluation (IME) will comprise a consultation with an independent general practitioner (IME GP) who will assess whether the sick listed worker has been given eligible and available opportunities in return to work follow-up in Norway. The independent medical evaluation general practitioner (IME GP) will write a short report that is sent to the treating general practitioner as input from a colleague. The report can be used in the follow-up of the sick listed participant. The participants in the treatment as usual (TAU) group will not receive any other follow-up than normal follow-up by the treating general practitioner. The qualitative evaluation will be conducted to gain insight into the experiences of the general practitioners and the participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants on sick leave with an International Classification of Primary Care-2 diagnosis will be recruited through the Norwegian Labour and Welfare Administration's (NAV) registries, when reaching 22 weeks of sick leave (full or graded).

Exclusion Criteria:

* People with International Classification of Disease-10 diagnoses, cancer or dementia.
* People who are pregnant.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7642 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in sick leave | Measured at three and eight weeks after randomization.
  Data on sickness benefits from official registers will be used to measure the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Silje Maeland, PhD, Principal Investigator — Uni Research Health
Locations (1):
- Uni Research, Bergen, Norway

REFERENCES:
- [Derived] Maeland S, Holmas TH, Oyeflaten I, Husabo E, Werner EL, Monstad K. What is the effect of independent medical evaluation on days on sickness benefits for long-term sick listed employees in Norway? A pragmatic randomised controlled trial, the NIME-trial. BMC Public Health. 2022 Feb 26;22(1):400. doi: 10.1186/s12889-022-12800-1. PMID 35216560
- [Derived] Oyeflaten I, Maeland S, Haukenes I. Independent medical evaluation of general practitioners' follow-up of sick-listed patients: a cross-sectional study in Norway. BMJ Open. 2020 Mar 18;10(3):e032776. doi: 10.1136/bmjopen-2019-032776. PMID 32193258
- [Derived] Aamland A, Husabo E, Maeland S. Independent medical evaluation for sick-listed patients: a focus group study of GPs expectations and experiences. BMC Health Serv Res. 2018 Aug 29;18(1):666. doi: 10.1186/s12913-018-3481-3. PMID 30157844
- [Derived] Husabo E, Monstad K, Holmas TH, Oyeflaten I, Werner EL, Maeland S. Protocol for the effect evaluation of independent medical evaluation after six months sick leave: a randomized controlled trial of independent medical evaluation versus treatment as usual in Norway. BMC Public Health. 2017 Jun 14;17(1):573. doi: 10.1186/s12889-017-4469-3. PMID 28615017